CLINICAL TRIAL: NCT02356172
Title: Psychological Outcomes in Isolated GNRH Deficiency
Status: Terminated | Type: Observational
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999915077; 15-CH-N077
Record Dates: First submitted 2015-02-04; First posted 2015-02-05 (Estimated); Last update posted 2019-07-18 (Actual); Status verified 2019-07-16

CONDITIONS: Hypogonadism
Keywords: Quality of Life; Depression; Kallmann Syndrome; Hypogonadotropic Hypogonadism
MeSH Terms: conditions — Hypogonadism; Depression; Kallmann Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional

GROUPS / COHORTS (2):
- Healthy Controls: Healthy males or females who are greater than or equal to 18 years old.
- Patients: Males or females with a diagnosis of IGD (Isolated GnRH Deficiency) who are greater than or equal to 18 years old.

SUMMARY:
Background:

- Isolated (or Congenital) GnRH Deficiency (IGD) is a rare disease. People who have this go through puberty late. Some never reach puberty or don t complete it without treatment. They also may have an impaired sense of smell or other health problems. Research shows that disorders like this can have a negative effect on a person s psychological profile.

Objective:

- To understand the psychological outcomes in people with IGD. These can include depression, anxiety, poor health, and poor social function.

Eligibility:

* Adults age 18 and over with IGD. They must be currently on a full dose of hormone replacement therapy for at least 3 months.
* Healthy adult volunteers.

Design:

* Participants will get a username and password. This will give them access to questions online. They can do this from any computer connected to the Internet.
* Participants will log in and complete the questionnaires. There are 5 total, but they will appear as 1 continuous set of questions. Answering them takes about 1 hour or less.
* The first set is about the participant s disorder. The rest ask about depression, anxiety, global health, and social function.
* All answers will be used for research and to better understand reproductive disorders. Only researchers from the NIH Unit on Genetics of Puberty and Reproduction and from this study will know which answers belong to which participant.

DETAILED DESCRIPTION:
Isolated GnRH Deficiency (IGD) is a rare disorder characterized by decreased secretion of GnRH, resulting in impaired gonadotropin secretion and subsequent impaired sex-steroid production. Patients with this rare clinical syndrome present with absent, delayed, or stalled pubertal development by eighteen years of age. In addition, non-reproductive phenotypes of this spectrum have been identified in some individuals, including anosmia, auditory and ocular defects, and skeletal, neurological, and renal anomalies.

Due to the complex heterogeneity among affected individuals and the rarity of the disease itself, the phenotypic spectrum has not been fully investigated. The relationship between psychological disorders and IGD remains largely unexplored as a phenotypic association, despite evidence that disorders of puberty and reproduction can have a negative impact on the psychological profile.

This study aims to conduct a preliminary investigation into the association between psychological symptoms and IGD. We plan to recruit adult patients with a diagnosis of IGD to complete online assessments that measure psychological health outcomes from the patient perspective in order to gauge the prevalence of negative emotional states among affected individuals, compared to healthy controls. This will determine whether further studies are necessary to investigate psychiatric disease as part of the phenotypic spectrum of the disorder, and will improve our understanding of this complex disorder as a whole. Greater knowledge of the psychological impact of IGD may impact the current standards of evaluation and treatment of patients with delayed pubertal maturation.

ELIGIBILITY:
* ELIGIBILITY CRITERIA FOR IGD PATIENTS:

INCLUSION CRITERIA:

Males or females with clinical findings consistent with IGD who are greater than or equal to 18 years old and treated with hormone replacement therapy for IGD at the full adult replacement dose for at least 3 months. Clinical findings of IGD will be confirmed by a nurse or physician associated with this protocol, and include: clinical presentation consistent with a diagnosis of IGD, such as delayed, incomplete, or absent pubertal development, and a record of serum hormone levels demonstrating low total testosterone (males) or estradiol (females) in association with low or inappropriately normal gonadotropin levels in a clinic note or history and physical, and individuals with records demonstrating failure to undergo normal puberty. Anosmia may or may not be present. Since IGD presents as a phenotypic spectrum, there are no specific exclusion criteria for this study, except as noted below.

EXCLUSION CRITERIA:

* Patients with a diagnosis of IGD who are <18 years old;
* Patients with a diagnosis of IGD who are not on a full adult replacement dose of sex hormone therapy for at least 3 months;
* Patients who do not have a diagnosis of IGD as indicated by the inclusion criteria above;
* Patients without access to a computer connected to the internet;
* Patients who cannot read, write, and understand English at an eighth grade level or above.

ELIGIBILITY CRITERIA FOR HEALTHY CONTROLS:

INCLUSION CRITERIA:

Healthy males or females who are greater than or equal to 18 years old.

EXCLUSION CRITERIA:

* Subjects with any chronic medical condition, other than seasonal/environmental allergies;
* Subjects with a BMI < 18.5 or > 29.9;
* Subjects with prior history of abnormal pubertal development, infertility, or anosmia;
* Subjects with a family history of IGD;
* Subjects without access to a computer connected to the internet;
* Subjects who cannot read, write, and understand English at an eighth grade level or above.

Ages: 18 Years to 200 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2015-02-04; Primary Completion 2017-06-01 (Actual); Study Completion 2019-07-16 (Actual)

PRIMARY OUTCOMES:
The primary outcome is to identify whether patients with Isolated GnRH Deficiency have a higher prevalence of negative emotional states, including depression, anxiety, poor social function and quality of life, than healthy controls. | At enrollment
  In analysis phase

CONTACTS AND LOCATIONS:
Overall Officials: Angela Delaney Freedman, M.D., Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (1):
- National Institute of Child Health and Human Development (NICHD), 9000 Rockville, Bethesda, Maryland, United States